CLINICAL TRIAL: NCT00677196
Title: The Canadian StoneBreakerTM Trial: A Randomized, Multicentre Trial Comparing The LMA StoneBreakerTM and the Swiss LithoClastR During Percutaneous Nephrolithotripsy.
Brief Title: The StoneBreakerTM Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: VGH and UBC Hospital Foundation (Other); Vancouver Coastal Health (Other Government)
Responsible Party: Dr. Ben Chew, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H07-01887
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2010-09-27 (Estimated); Status verified 2010-09

CONDITIONS: Percutaneous Nephrolithotripsy
Keywords: PNL; Lithoclast; Stonebreaker; efficiency stone fragmentation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): The LMA StoneBreakerTM
  Interventions: Device: The stonebreaker arm (LMA Stonebreaker)
- 2 (Active Comparator): Pneumatic Lithotripsy
  Interventions: Device: Pneumatic Lithotripsy (Swiss LithoClastR)

INTERVENTIONS:
Device: The stonebreaker arm (LMA Stonebreaker) — The interventional device name is the LMA Stonebreaker pneumatic handheld lithotriptor.
  Arms: 1
Device: Pneumatic Lithotripsy (Swiss LithoClastR) — Pneumatic lithotripsy, the Swiss LithoClastR during percutaneous nephrolithotripsy (PNL)
  Arms: 2

SUMMARY:
The purpose of this study is to compare the LMA StoneBreakerTM to the current standard of pneumatic lithotripsy, the Swiss LithoClastR, during percutaneous nephrolithotripsy (PNL).

DETAILED DESCRIPTION:
Objective:

The purpose of this study is to compare the LMA StoneBreakerTM to the current standard of pneumatic lithotripsy, the Swiss LithoClastR, during percutaneous nephrolithotripsy (PNL).

Rationale:

Percutaneous nephrolithotripsy (PNL) is the preferred treatment modality for renal stones greater than 2cm in diameter.

The pneumatic lithotriptor functions as a pneumatic jackhammer, providing either a single pulse or a train of pulses at 2Hz as determined by the operator. Its chief advantage is its ability to fragment even the hardest calculi. The pneumatic lithotriptor, while extremely effective, does not utilize thermal energy and therefore has no risk of thermal damage to the surrounding tissue. The pneumatic lithotriptor currently in use, the Swiss LithoClast is powered by compressed medical air. The primary disadvantage of this device is that the residual calculi must be individually removed with forceps following fragmentation.

The StoneBreaker, manufactured by the Laryngeal Mask Airway Company, is a novel hand-held pneumatic lithotriptor. This device is powered by a compressed carbon dioxide cartridge.

Hypothesis:

The LMA StoneBreaker, provides more efficient lithotripsy of renal calculi treated by PNL over the existing pneumatic intracorporeal lithotriptor the Swiss LithoClast.

Methods:

Patients would be recruited to the study from the clinical population who present for stone management at VGH. None of the physicians involved has a financial interest in either of the devices being evaluated. The purpose is to compare the pneumatic lithotripsy devices and is not an evaluation of PNL, a procedure whose safety and efficacy is well established.

Patients who consented to PNL for management of their renal stone would be approached about entry into the study by either of the primary surgeons, the research coordinator, or the research fellows. Patients would understand that PNL is not an experimental procedure and that the research project specifically is comparing the two lithotripsy devices with similar mechanism of action and safety profile. The goal in all cases would be to render the patient stone free. The patients care would not deviate from our standard PNL care protocol, summarized below, with the exception of the use of a different lithoclast.

Pre-operatively, the patients are assessed in the Preanaesthetic clinic as necessary. Blood tests including CBC and differential, blood type and antibody screen, creatinine and electrolytes are routinely obtained. Urine samples will be sent preoperatively for culture and sensitivity. If the urine culture is positive, organism specific antibiotics will be prescribed prior to treatment. If the urine culture is negative, prophylactic antibiotics will be ordered and administered, prior to the induction of anaesthesia, by the treating surgeon.

Our standard operative protocol for PNL as described next will be followed for all cases. After receiving a general anaesthetic, cystoscopy and placement of a ureteral catheter on the affected side may be performed. The will be used to perform retrograde pyelography in order to determine the optimal access site to the kidney. A Foley catheter will be placed to drain the bladder throughout the procedure. Next, under fluoroscopic guidance, access to the affected renal collecting system will be obtained with a needle down which a guide wire is passed by the interventional radiology department or the operating surgeon.

The tract will be dilated to accommodate the 30F working sheath. The stone will then be visualized and fragmented with either of the two devices, determined by randomization. Remaining fragments will be removed using grasping forceps and an ultrasound suction device until the patient is rendered stone free. A final visual inspection of the collecting system will ensure the patient is stone free. The choice of renal drainage method after the procedure will be left to the discretion of the treating surgeon.

Statistical Analysis: Student's t-test and ANOVA will be used to determine statistical significance. P-values < 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 undergoing PNL
* Previously untreated renal stones
* Patients with 3 or less individual renal calculi, accessible with a rigid nephroscope
* Stones must be at least >225mm2 area on KUB
* Patient must have a CT scan prior to treatment

Exclusion Criteria:

* Patients with an active contraindication for PNL (pregnancy, uncorrected coagulopathy, active urinary infection, contrast allergy)
* Partial staghorn calculi
* Complete staghorn calculi
* Stones in calyceal diverticulum
* Cases requiring multiple tracts

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Time to complete fragmentation of renal calculi treated via PNL | During surgery

SECONDARY OUTCOMES:
Time to removal of large fragments using graspers & time required with US to remove small fragments/dust | During surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ben Chew, MD, FRCSC, Principal Investigator — University of British Columbia; R. Paterson, MD, Study Director — University of British Columbia; J. Wright, MD, Study Director — University of British Columbia; J. Teichman, MD, Study Director — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada